CLINICAL TRIAL: NCT05318469
Title: A Phase I/II Study Evaluating the Safety and Efficacy of Ivermectin in Combination With Immune Checkpoint Inhibitor in Patients With Metastatic Triple Negative Breast Cancer
Brief Title: Ivermectin in Combination With Balstilimab or Pembrolizumab in Patients With Metastatic Triple Negative Breast Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yuan Yuan (Other)
Collaborators: Agenus Inc. (Industry); Gateway for Cancer Research (Other)
Responsible Party: Sponsor-Investigator, Yuan Yuan, Medical Director, Breast Oncology DRG, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022-07-YUAN-IB-TNBC
Record Dates: First submitted 2022-04-01; First posted 2022-04-08 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Ivermectin; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ivermectin, balstilimab) (Experimental): Patients will receive balstilimab 450 mg or pembrolizumab 200 mg, IV, on Day 1 of each 3 week cycle and ivermectin at the assigned dose (see Section 5.1, Table 5.1.2), PO, Days 1-3, 8-10, 15-17 of each cycle (Days 1-3 of each week) until disease progression, intolerable toxicities, withdrawal of consent, or up to 35 treatments or 2 years of balstilimab or pembrolizumab, whichever comes first
  Interventions: Drug: Ivermectin; Drug: Balstilmab; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Ivermectin — Ivermectin at the assigned dose administered PO on Days 1-3, 8-10, 15-17 of each 21 day cycle (Days1-3 of each week).
  Other Names: Sklice; Stromectol
Drug: Balstilmab — Balstilimab 300 mg administered intravenously on Day 1 of each 21 day cycle.
Drug: Pembrolizumab — Pembrolizumab 200 mg IV on Day 1 of each 21 day cycle

SUMMARY:
This phase II trial studies the side effects and best dose of ivermectin in combination with balstilimab or pembrolizumab and to see how well they they work in shrinking tumors in patients with triple negative breast cancer that has spread to other places in the body (metastatic). Immunotherapy with monoclonal antibodies, such as balstilimab or pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Ivermectin may help block the formation of growths that may become cancer. Giving ivermectin with balstilimab or pembrolizumab may increase the effect of balstilimab or pembrolizumab in shrinking tumors in patients with triple negative breast cancer. The secondary objectives of the study include evaluating the following efficacy outcomes: objective response rate (ORR), progression free survival (PFS), overall survival (OS), duration of response (DOR), clinical benefit rate (CBR), and patients' quality of life (QOL) by European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30).

DETAILED DESCRIPTION:
Patients receive ivermectin orally (PO) once daily (QD) on days 1-3, 8-10, and 15-17. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also receive balstilimab or pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 21 days for up to 35 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 90 days and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) ≤ 1
* Life expectancy > 3 months
* Histologically confirmed metastatic triple negative breast cancer. Triple negative status will be defined as estrogen receptor (ER) and progesterone receptor (PR) ≤ 10% and HER2 negative (by immunohistochemistry [IHC] or fluorescence in situ hybridization [FISH]), per American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines
* Patients must have progressed on 1-2 prior lines of systemic therapy (chemotherapy and/or drug-antibody conjugate) in the metastatic setting
* Measurable or evaluable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
* Fully recovered from the acute toxic effects (except alopecia) to ≤ grade 2 from prior anti-cancer therapy
* For Phase 2 expansion only, must be PD-L1 negative. Note: For Phase 1 safety cohort, any PD-L1 status will be allowed to enroll.
* Patients must have adequate organ function as defined in the following:
* Absolute neutrophil count (ANC) ≥ 1,500/mm^3
* Platelets ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL or ≥ 5.6 mmol/L. Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks
* Total serum bilirubin ≤ 1.5 x upper limit of normal (ULN) OR direct bilirubin ≤ ULN for participants with total bilirubin levels > 1.5 x ULN
* Aspartate aminotransferase (AST) ≤ 1.5 x ULN or ≤ 3 x ULN with liver metastases
* Alanine aminotransferase (ALT) ≤ 1.5 x ULN or ≤ 3 x ULN with liver metastases
* Creatinine ≤ 1.5 x ULN OR calculated creatinine clearance ≥ 30 mL/min for participant with creatinine levels >1.5 x institutional ULN
* International normalized ratio (INR) or prothrombin time (PT), activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
* Left ventricular ejection fraction (LVEF) ≥ 50% by echocardiogram
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* A male participant must agree to use a contraception during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * Females of child-bearing potential must be willing to use effective contraception during study and for 120 days after the last dose
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
* Prohibited Treatments and/or Therapies:
* Chemotherapy, radiation therapy, biological therapy, immunotherapy within 28 days prior to day 1 of protocol therapy
* Prior immune checkpoint inhibitor therapy in metastatic setting (Note: Prior use of immune checkpoint inhibitor in neoadjuvant or adjuvant setting only permitted if last dose is at least 1 year from start of study intervention)
* Prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease
* Any live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed
* Participants on any dose of warfarin. Use of low molecular weight heparin, antithrombin agents, anti-platelet agents or factor Xa inhibitors is allowed
* Participants may not be currently participating in or participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention
* Issues with tolerating oral medication (e.g., inability to swallow pills, malabsorption issues, ongoing nausea or vomiting during screening)
* Women who are or are planning to become pregnant or breastfeed
* Known allergy to any of the components within the study agents and/or their excipients
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for at least three years
* Participants must not have known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention
* History of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Active infection requiring systemic therapy
* Known history of Human Immunodeficiency Virus (HIV) infection
* Known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority
* Known history of active TB (Mycobacterium tuberculosis)
* Intercurrent or historic medical condition that increases subject risk in the opinion of the Investigator. Eligibility may be revisited for intercurrent medical conditions once resolution/recovery is deemed adequate by the investigator (e.g., recovery from major surgery, completion of treatment for severe infection).
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment
* Has had an allogenic tissue/solid organ transplant
* Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) class II, unstable angina, myocardial infarction, or stroke within 6 months of the first dose of study drug, or cardiac arrhythmia requiring medical treatment at screening
* Subjects having > 1+ proteinuria on urine dipstick testing unless a 24-hour urine collection for quantitative assessment indicates that the urine protein is < 1 g/24 hours
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-10-13 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | From start of study treatment until 90 days after treatment completion
  Phase 1: To determine the recommended phase 2 dose of ivermectin in combination with balstilimab or pembrolizumab using NCI-CTCAE v5.0
Objective response rate | From start of study treatment until disease progression, intolerable toxicities, or withdrawal of consent. Assessed up to 2 years.
  Phase 2: To determine the efficacy of ivermectin in combination with balstilimab or pembrolizumab in mTNBC using the objective response rate (ORR)

SECONDARY OUTCOMES:
Objective response rate | From start of study treatment until disease progression, intolerable toxicities, or withdrawal of consent. Assessed up to 2 years.
  Evaluate the efficacy of ivermectin in combination with balstilimab or pembrolizumab in mTNBC using objective response rate (ORR) using RECIST 1.1
Progression free survival | From start of study treatment until disease progression, intolerable toxicities, or withdrawal of consent. Assessed up to 6 years.
  From start of therapy until first documentation of disease progression per RECIST 1.1 or death due to any cause.
Overall survival | From start of study treatment to death or last contact. Assessed up to 6 years
  From start of study treatment to date of death due to any cause. Patient's last known to be alive are censored at date of last contact.
Duration of response | From the date of first objective response recorded until disease progression, death or last contact. Assessed up to 6 years
  Measured from the date of first objective response recorded (CR or PR) until progression per RECIST 1.1, death or last contact (censored). Patient's last known to be alive are censored at date of last contact.
Clinical benefit rate | From start of study treatment until disease progression, intolerable toxicities, or withdrawal of consent. Assessed up to 6 years.
  Defined as progression-free for at least 6 months or CR or PR per RECIST 1.1.
Patients' quality of life | On day 1 of each 3 week cycle and at end of treatment visit. Assessed up to 2 years.
  Evaluated by European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30) version 3.0 per standardized EORTC scoring guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Yuan, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States